CLINICAL TRIAL: NCT06440512
Title: The Effect of Chocolate on Vascular Function of Endurance Runners
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Evangelia Kouidi, Professor, Director of the Laboratory of Sports Medicine, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: EC-161/2023
Record Dates: First submitted 2024-05-22; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Vascular Function
Keywords: arterial stiffness; aerobic fitness; chocolate; polyphenols; endurance runners

STUDY DESIGN:
Intervention Model Description: This study employs a crossover design to investigate the effects of chocolate consumption on vascular function of endurance runners. Participants will undergo multiple treatment periods where they will receive either dark chocolate or white chocolate, followed by washout periods to minimize carryover effects. The order of treatment administration will be randomized to mitigate potential sequence effects. Outcome measures will be assessed at the end of each treatment period to evaluate the impact of chocolate consumption on vascular function, athletic performance and other relevant outcomes.
Masking Description: Τhe study does not use the method of blind evaluation due to the nature of the interventions, which are easily identifiable by the participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A Chocolate Arm (Experimental): Intervention period 1:The group will consume 50 grams of dark chocolate daily for two weeks.
  Washout period: Two-weeks
  Intervention period 2: The group will consume 40 grams of white chocolate daily for two weeks.
  Interventions: Other: Dark chocolate Intervention; Other: White chocolate Intervention
- B Chocolate Arm (Experimental): Intervention period 1:The group will consume 40 grams of white chocolate daily for two weeks.
  Washout period: Two-weeks
  Intervention period 2: The group will consume 50 grams of dark chocolate daily for two weeks
  Interventions: Other: Dark chocolate Intervention; Other: White chocolate Intervention

INTERVENTIONS:
Other: Dark chocolate Intervention — The intervention involves daily consumption of 50 grams of dark chocolate for a period of two weeks. The dark chocolate is provided in tablet form, and participants are instructed to consume it daily.
Other: White chocolate Intervention — The intervention involves daily consumption of 40 grams of white chocolate for a period of two weeks. The dark chocolate is provided in tablet form, and participants are instructed to consume it daily.

SUMMARY:
The aim of this study is to examine the effects of chocolate on the vascular function of endurance runners through a crossover study involving male runners consuming both dark and white chocolate.

DETAILED DESCRIPTION:
Participants will be male endurance runners who will receive both black and white chocolate interventions. Arterial stiffness, cardiovascular parameters, respiratory parameters, and running performance will be assessed before and after each intervention period. The study will involve a two-week intervention period for each type of chocolate, with a washout period in between. The primary outcome measure will be arterial stiffness, while secondary outcome measures will include cardiovascular and respiratory parameters, as well as running performance. The study is expected to provide insights into the effects of chocolate consumption on vascular function in endurance athletes.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Male
* Age: 25-55 years
* Healthy status
* Active endurance runner
* Regular physical activity (at least 3 times per week)
* Availability on specific days and times for research sessions
* Willingness and consistency

Exclusion Criteria:

* Allergies or Intolerances: Participants with known allergies or intolerances to chocolate or any of its ingredients.
* Cardiovascular Diseases: Participants with known cardiovascular diseases or history of cardiac episodes.
* Metabolic Disorders: Individuals with diabetes or other metabolic disorders that may affect glucose and insulin metabolism.
* Contradictory Diet: Individuals following specific diets that may affect the study, such as high or low flavonoid diets.
* Medication Use: Individuals taking medications that affect vascular function, such as antihypertensives or anticoagulants.
* Smoking: Smokers or individuals who have quit smoking within the last six months.
* Substance Abuse: Individuals with a history of alcohol or substance abuse.
* Patients with Chronic Diseases: Individuals with serious chronic diseases that may affect the study outcomes.
* Participation in Other Studies: Individuals participating in other clinical trials or research that may affect the study outcomes.
* Physical Condition: Individuals who are not regular runners or who do not exercise regularly at a level similar to other participants.

Ages: 25 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-10 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-11-20 (Estimated)

PRIMARY OUTCOMES:
CF-PWV (Carotid-Femoral Pulse Wave Velocity) | Baseline and at the end of each 2-week intervention period (after consumption of dark chocolate and after consumption of white chocolate).
  Measurement of the velocity of the pressure wave between the carotid and femoral arteries, expressed in meters per second (m/s)
AIx (Augmentation Index) | Baseline and at the end of each 2-week intervention period (after consumption of dark chocolate and after consumption of white chocolate).
  Measurement of arterial stiffness, calculated as the difference between the first and second systolic peaks of the arterial waveform, expressed as a percentage (%)
Exercise Time in Cardiopulmonary Exercise Testing | Baseline and at the end of each 2-week intervention period (after consumption of dark chocolate and after consumption of white chocolate).
  Total duration of exercise during cardiopulmonary exercise testing, measured in minutes.
VO2max (Maximal Oxygen Uptake) | Baseline and at the end of each 2-week intervention period (after consumption of dark chocolate and after consumption of white chocolate).
  Maximum amount of oxygen consumed per minute during incremental exercise, expressed in milliliters per kilogram per minute (mL/kg/min)
5km Time | Baseline and at the end of each 2-week intervention period (after consumption of dark chocolate and after consumption of white chocolate).
  Total time taken to complete a 5-kilometer run, measured in minutes and seconds.
5km Speed | Baseline and at the end of each 2-week intervention period (after consumption of dark chocolate and after consumption of white chocolate).
  Average speed during a 5-kilometer run, expressed in kilometers per hour (km/h).

CONTACTS AND LOCATIONS:
Overall Officials: Evangelia Kouidi, Professor, Principal Investigator — Aristotle University Of Thessaloniki
Locations (1):
- Laboratory of Sports Medicine, Thessaloniki, Greece